CLINICAL TRIAL: NCT04745156
Title: Inducing Functional Plasticity in Glioma-Involved Functional Cortex With Deficit-Inducing Cortical Stimulation and Targeted Behavioral Therapy to Increase Extent of Resection
Brief Title: A Study Using Brain Stimulation and Behavioral Therapy to Increase Extent of Resection in Low-Grade Gliomas
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Max Krucoff, MD, Assistant Professor of Neurological Surgery, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PRO00039766
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Glioma; Glioma Intracranial; Gliomas Benign; Brain Tumor; Brain Cancer; Motor Cortex; Lesion
Keywords: Brain Stimulation; NeuroPace; Cortex Stimulation; Neuroplasticity; Plasticity; Hand Motor Cortex; Primary Motor Cortex; M1; Motor Mapping; Resection; Surgery; Motor Rehabilitation; Prehabilitation
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- RNS System Implantation (Experimental): This is a device feasibility study, therefore participants will only be enrolled into the investigational arm and will receive the RNS System Implantation.
  Interventions: Device: RNS System Implantation

INTERVENTIONS:
Device: RNS System Implantation — Following resection consistent with SoC, if there is evidence of residual tumor which cannot be resected due to invasion of hand-M1 but which is small enough to be covered by two four-electrode strips, these strips will be placed on the functional cortex of interest and secured to the dura. The location of the leads will be registered into the navigation software (either Medtronic Stealth or Brainlab). The dura will then be closed as watertight as possible, and the RNS System will be incorporated into the craniotomy on closure Prior to closure, four bone screws will be placed and registered to the intraoperative navigation system as internal fiducials to be retrieved for future procedures.

SUMMARY:
This study uses a cranial implant to deliver cortical stimulation that, when paired with physiotherapy, will remap the brain so that critical brain functions can be protected during brain tumor surgery. This pilot study will provide initial evidence for the safety and feasibility of such a protocol which will lead to future pivotal trials that could radically change eloquent area brain surgery. For patients with otherwise incompletely resectable brain tumors, this could mean a longer life expectancy and a better quality of life.

DETAILED DESCRIPTION:
Study Protocol: Participants will undergo a standard-of-care craniotomy for resection of low-grade glioma. If part of the lesion cannot be removed due to involvement of functional cortex, RNS (Responsive Neurostimulation System [RNS; NeuroPace, Inc.]) electrodes will be implanted over the tumor-invaded area(s) in five participants. Stimulation will then be optimized for each individual to disrupt the function of the invaded cortical node (e.g., hand motor area -> hand dysfunction) (Aim 1). Over the next two months, outpatient physiotherapy will work to overcome the stim-induced deficits through gradual increases in stimulation amplitude as other, non-stimulated brain regions begin to assume its function (Aim 2). Once complete, participants will return to the OR for device explantation, repeated intraoperative mapping, and extended resection (if safe) (Aim 3).

Aim 1: Optimize stimulation to maximize stim-induced deficits and minimize side effects Rationale: To induce plasticity, stimulation parameters must be individually tuned to maximize effect and minimize side effects. Approach: After device implantation and prior to hospital discharge, stimulus settings (frequency, pulse-width, and amplitude) will be optimized to the relevant clinical response while minimizing adverse effects (e.g., focal tonus, myoclonus, or seizures) while still in the safe, inpatient setting. Outcomes: Primary Endpoints: 1) stim-induced focal clinical deficit as measured on the relevant clinical scale (e.g., manual motor score [0-5], picture naming [x/10]), repetition [x/3]); 2) stim-induced side effects (e.g., seizures).

Aim 2: Evaluate extent of remapping and safety of outpatient stimulation-physiotherapy protocol. Rationale: The ability to deliver chronic, outpatient stimulation is vital for practical clinical translation, yet neither its safety nor efficacy has been demonstrated. Approach: After Aim 1, a physiotherapist will assign a personalized, outpatient therapy regimen aimed at overcoming stim-induced deficits. Participants will have daily virtual sessions and return to clinic 2x/week for amplitude increases to re-induce deficits that therapy has overcome. This will continue until stimulation no longer can induce a deficit, suggesting successful functional remapping and enabling a return to the OR for further resection. Outcomes: Primary Endpoints: 1) absence of stim-related ER visits, readmissions, or serious adverse events (safety), 2) changes in intraop stimulation maps from surgery 1 to surgery 2 (induced remapping).

Aim 3: Evaluate ability to extend surgical resections and associated neurological outcomes. Rationale: Any change in functional boundaries will only be useful if it results in a safe, extended resection. Approach: Each surgery will proceed with standard-of-care intraoperative functional mapping techniques and decision making. Neurological examinations will be performed preoperatively, daily while inpatient, then again at 2-weeks and 3-months postoperatively. Extent of resection will be evaluated as 3D residual tumor volume on postoperative MRI. Outcomes: Primary Endpoint: 1) Change in residual tumor volume after second versus first resection, 2) new neurological deficits 3-months after second resection compared to before second resection. Secondary Endpoint: 1) New, temporary neurological deficits after the second surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. Ability to understand a written informed consent document, and the willingness to sign it
3. Radiographic evidence of likely low-grade glioma on MRI (i.e. non-enhancing) invading primary motor cortex in the non-dominant hemisphere.
4. Karnofsky performance status (KPS) ≥ 75
5. Normal or near normal motor strength (i.e., at least 3/5 in relevant areas)
6. Normal or near normal speech (Can consistently name at least 4/5 cards)
7. No medical contraindication to surgery
8. Free of other illness that may shorten life expectancy

Exclusion Criteria:

1. Presence of other malignancy not in remission
2. Evidence of bi-hemispheric or widespread tumor involvement
3. Likely candidate to receive GTR on initial resection
4. Medically high-risk surgical candidate
5. History of recent scalp or systemic infection
6. Presence of other implants or foreign bodies in the head
7. Inability to receive an MRI for any reason
8. Inability to receive cortical stimulation for any reason
9. Coagulation disorders and/or use of anti-thrombotic therapies
10. Platelet count < 50
11. Diathermy procedures
12. Electroconvulsive Therapy (ECT)
13. Transcranial Magnetic Stimulation (TMS)
14. Presence of implanted cardiac device (such as a pacemaker or defibrillator)
15. Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Extent of resection | Within 1 week after second surgery
  Calculated as: Tumor volume after second surgery - tumor volume before second surgery. Determination of volumes will be made by an attending radiologist without knowledge of clinical outcome. Manual segmentation will be performed to measure tumor volumes based on fluid-attenuated inversion recovery (FLAIR) axial slices.
Stimulation-induced motor deficits | Within 2 weeks after first surgery
  Calculated as manual muscle score (MMS) before stimulation - MMS after stimulation.
  MMS is a zero-to-five scale assessed as the following:
  5 - normal strength 4 - give away weakness 3 - movement against gravity 2 - movement in anti-gravity position
  1 - muscle twitch 0 - no movement
Stimulation-induced language deficits | Within 2 weeks after first surgery
  3a. Calculated as picture naming score (x/10) before stimulation minus after stimulation.
  3b. Calculated as sentence repitition score (x/3) before stimulation minus after stimulation.
Stimulation-induced side effects | Within 2 weeks after first surgery
  Reported as number of unintended stimulation effects, such as myoclonus, tonus, seizures, or unpleasant sensations
Safety of outpatient stimulation-therapy protocol | Up to 8 weeks
  Reported as number of stimulation- or physiotherapy related ER visits, readmissions, or serious adverse events
Stimulation-induced brain remapping | This data will be obtained intraoperatively during the second surgery
  This outcome will be reported as a descriptive variable, calculated as changes in the intraoperative stimulation map obtained during surgery 2 compared to surgery 1
Number of participants with a new neurological deficit | Assessed at 3-month postoperative visit after second surgery
  Any new, permanent neurological deficits resulting from the second surgery

CONTACTS AND LOCATIONS:
Overall Officials: Max Krucoff, MD, Principal Investigator — Medical College of Wisconsin